CLINICAL TRIAL: NCT06306235
Title: Are Non-participants of Conventional Centre-based Cardiac Rehabilitation Willing to Participate in Cardiac Telerehabilitation?
Status: Completed | Type: Observational
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20.84-reva20.06
Record Dates: First submitted 2020-10-12; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2022-10

CONDITIONS: Cardiac Rehabilitation
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Part A: 30 patients will be interviewed. Part B: 300 patients will complete written questionnaire on tablet.

SUMMARY:
Patients who are eligible for cardiac rehabilitation but do not want to participate will be offered to participate in an interview (part A of the study) or a tablet questionnaire (part B of the study).

Goal is to identify main barriers for conventional rehabilitation as well as to assess willingness to participate in cardiac telerehabilitation, main barriers and willingness-to-pay for cardiac telerehabilitation.

DETAILED DESCRIPTION:
Cardiac rehabilitation (CR) is indicated in patients with a wide range of cardiovascular diseases. Its benefits are well-studied and participation in CR is thus stated as a Class IA recommendation in the 2016 European Guidelines on cardiovascular disease prevention in clinical practice. It is known however that participation rates are low. This is due to multiple factors such as health system barriers (e.g. lack of referral by doctors), as well as patient factors (eg. travelling time to hospital).

Telerehabilitation is a modality of cardiac rehabilitation that is widely studied to overcome barriers in conventional cardiac rehabilitation. Most studies about telerehabilitation screen for potential rehabilitation candidates, ask which patients are prepared to start centre-based rehabilitation and then start randomisation for centre-based or home-based rehabilitation.

The hypothesis is that by offering a home-based alternative for centre-based rehabilitation, patient participation rates will go up. However, this hypothesis has not been investigated.

The willingness to participate in patients that refuse centre-based rehabilitation is thus scarcely studied.

This study aims to assess the willingness to participate in telerehabilitation in patients that refuse conventional centre-based rehabilitation as well as the main reasons not to participate in centre-based rehabilitation.

Methods

Patients that are eligible for participating in cardiac rehabilitation will be offered to do so as usual. Those who do not wish to participate or are not sure whether they will participate in cardiac rehabilitation will be asked to participate in this study.

The first part of this study is a pilot part in which 30 patients will be included. These patients will be interviewed by one of the researchers (dr. Maarten Falter or dr. Martijn Scherrenberg). A semi-structured interview of 20 minutes will be performed to assess the most important barriers for rehabilitation, willingness-to-pay and possible barriers for telerehabilitation, as well as patient profile and socio-economic background. Informed consent will also be asked to collect patient data from the hospital records (age, gender, cardiac disease, cardiac index event, cardiac device implanted, indication for rehabilitation, date of primary cardiac event, length of hospital stay, cardiac rehabilitation history, procedures performed, comorbidities, distance from home to hospital, Mobiscore, smoking status, length, weight, medication, ejection fraction) as these factors are possible determinants of the outcome of our study.

The second part of this study is a survey that will assess the most important barriers in 300 patients. This survey will be constructed using the main barriers found in literature in combination with main barriers mentioned by the pilot population. The survey will consist of multiple-choice questions and will again assess main barriers for participating in rehabilitation and telerehabilitation. The survey will be completed using an iPad from the cardiology department using Qualtrics while the patient is still in the hospital. The Qualtrics license is obtained via Hasselt University. Informed consent will also be asked to collect patient data from the hospital records (see variables above).

All study results will be stored on a secured drive of Jessa hospital (K-drive). Only the health professionals with a therapeutic relation, the principal investigator and the local investigator can access this list. Data will be converted into a pseudonymized database for further statistical analysis in collaboration with the University of Hasselt or for analysis in collaboration with bachelor students of the University of Hasselt. Patients will only be included in the Jessa hospital.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for conventional cardiac rehabilitation
* Not willing to participate in conventional cardiac rehabilitation.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that are eligible for participating in cardiac rehabilitation will be offered to do so as usual. Those who do not wish to participate or are not sure whether they will participate in cardiac rehabilitation will be asked to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Willingness to participate in telerehabilitation | Immediate assessment of willingness during patient interview.
  Is the patient willing to participate in telerehabilitation? Based on question asked in interview, response will be recorded and evaluated by two independent investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Dendale, Principal Investigator — Jessa Hospital
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will not be shared. Pseudonymized data might be used for statistical support.